CLINICAL TRIAL: NCT06390358
Title: Acute and Chronic Effects of Tefillin Use on Remote Cardiac Ischemic Preconditioning
Brief Title: Effects of Remote Cardiac Ischemic Preconditioning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jack Rubinstein (Other)
Responsible Party: Sponsor-Investigator, Jack Rubinstein, Professor of Medicine, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-0733
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Function and Preconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tefillin (Experimental): Wearing of tefillin in traditional manner
  Interventions: Other: Tefillin
- Capsaicin (Active Comparator): Applying cream to non-dominant arm
  Interventions: Other: Tefillin

INTERVENTIONS:
Other: Tefillin — Wrapping of arm

SUMMARY:
A heart attack occurs when blood flow is disrupted to the heart and is related to both the blockage and flow restoration (reperfusion injury). An occlusion during a heart attack can be cleared (mostly via stents), but there are no methods to decrease reperfusion injury even though animal studies have found that "preconditioning" has powerful protective effects. Through the observation of Jewish men wearing tefillin the investigators have discovered a method of bringing preconditioning to patients at risk for heart attacks. This study will focus on women as the majority of people who wear tefillin (and have been studied) are men.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) is a process via which short bursts of ischemia result in dramatic subsequent protection in remote organs from a prolonged ischemic injury such as myocardial infarction from reperfusion injury. The translation of RIPC stimuli to clinically relevant therapies has not been successful as almost all prior research on RIPC (animal and human) involved the full blockage of blood flow to an organ or extremity (in humans commonly with full inflation cycles of a blood pressure cuff). Our laboratory's key translational insight involved the Jewish tradition of donning tefillin (phylacteries) that is traditionally worn on an almost daily basis by Jewish orthodox men on the non-dominant arm in a non-obstructive manner (NOB).

My laboratory has made substantial progress by demonstrating that tefillin induced NOB induces an RIPC phenotype in healthy (mostly) men. The overarching hypothesis of this proposal is that full arm NOB via tefillin results in a preconditioning stimulus in women that is sufficient to induce an RIPC phenotype. The sole aim will test the hypothesis that full arm NOB (in healthy females) results in an inducible RIPC phenotype that increases over time as measured via clinically relevant variables derived from heart rate variability monitoring and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Females over 18 years of age

Exclusion Criteria:

* Current medication use for medical condition or active medical condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified females
Enrollment: 24 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | 6 days
  HRV is determined by measuring the beat-to beat intervals.

SECONDARY OUTCOMES:
Inflammatory changes | 6 days
  Plasma will be analyzed for CCR2, CX3CR1, MCP-1 and VCAM1 and monocytes will be analyzed via migration and adhesion assays.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No